CLINICAL TRIAL: NCT03073174
Title: Dietary Intakes and Periodontal Outcomes After Sanative Therapy: A Follow-Up Study
Brief Title: Dietary Intakes and Periodontal Health: A Follow-Up Study
Status: Completed | Type: Observational
Sponsor: Brock University (Other)
Collaborators: Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery (Other)
Responsible Party: Principal Investigator, Wendy E. Ward, Ph.D., Professor and Canada Research Chair, Brock University
Other Study IDs: 16-131
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Periodontal Attachment Loss; Periodontal Pocket
Keywords: dietary intake; nutritional supplements; sanative therapy; healing; flavonoids; tea
MeSH Terms: conditions — Periodontal Attachment Loss; Periodontal Pocket

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva is being collected at time of hygiene appointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A previous study, on which this study is based, found that a diet higher in fruits and vegetables, beta-carotene, vitamin C, alpha-tocopherol, and fish oils (specifically eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA)) was positively associated with periodontal healing after sanative therapy (NCT02291835). The investigator's next step, in the present study, is to determine long-term benefits of sanative therapy in which patients have regular maintenance hygiene cleanings on periodontal health. Specifically, the relationship between intakes of specific foods, nutrients and supplements with clinical periodontal outcomes will be studied.

DETAILED DESCRIPTION:
Periodontitis is a chronic oral infection that results in the breakdown of connective tissue and alveolar bone that support the teeth. Bacteria and the body's own immune system mediate the severity of periodontitis, where teeth may become loose, fall out or have to be removed. Sanative therapy is a non-surgical process involving mechanical debridement of bacterial biofilms on roots of teeth, below the gum line. Participants in this present study previously underwent sanative therapy several years ago and have been attending the clinic for regular maintenance appointments to maintain periodontal health. While significant associations were observed with higher intakes of fruits and vegetables and specific nutrients (vitamins C and E, beta-carotene, fish oils) within a few months after sanative therapy, this study will follow-up these findings to determine if such relationships persist during a period of relatively stable periodontal health. Given new insights into a potential role of flavonoids in maintaining periodontal health, this aspect will also be studied. The overall objective is to determine if higher intakes of foods, nutrients and supplements known to have osteogenic and immunomodulatory effects are associated with improved clinical outcomes in individuals who previously underwent sanative therapy. At the regular maintenance appointment, clinical measures will be evaluated (clinical attachment loss, probing depth, bleeding on probing, plaque index). As well, the following will be evaluated: dietary intakes of macronutrients and micronutrients using the Block 2015 food frequency questionnaire; intakes of fruit, vegetables and fiber using the Block Dietary Fruit-Vegetable-Fiber Screener; nutritional supplement use and tea intake using specially developed questionnaires and salivary markers of inflammation using biochemical assays.

ELIGIBILITY:
Inclusion Criteria:

* previously participated in the original study (NCT02291835)

Exclusion Criteria:

* under 19 years of age
* have not participated in the previous study as this study is a direct follow-up of those participants

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who previously underwent sanative therapy to manage periodontal disease and who have regular maintenance periodontal cleanings on a regular basis at the clinic.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Loss (CAL) (also called Periodontal Attachment Loss) | At maintenance appointment (1 hour)
  Clinical Attachment Loss is a routine clinical measure of periodontal health (measured in mm)

SECONDARY OUTCOMES:
Probing Depth | At maintenance appointment (1 hour)
  Probing depth is a routine clinical measure of periodontal health (measured in mm)
Bleeding on Probing | At maintenance appointment (1 hour)
  Bleeding on Probing is a measure of inflammation and determined as the percent of bleeding sites that are measured at 6 sites per tooth.
Plaque Index | At maintenance appointment (1 hour)
  O'Leary Plaque Score Index is a score of the total amount of plaque present at 4 surfaces of the tooth.

OTHER OUTCOMES:
Dietary Nutrient Intakes | At maintenance appointment (1 hour)
  Dietary intakes measured using the Block food frequency questionnaire
Tea Intakes | At maintenance appointment (1 hour)
  Quantity and type of tea consumed will be determined using a questionnaire
Servings of Fruits, Vegetables and Fiber | At maintenance appointment (1 hour)
  A questionnaire called the Block Fruit-Vegtable-Fiber Screener is used to provide a score that pertains to number of servings of fruits, vegetables and fiber consumed over past month
Dietary Supplement Intakes | At maintenance appointment (1 hour)
  Intakes of specific dietary supplements measured using a dietary supplement questionnaire
Salivary Markers of Inflammation | At maintenance appointment (1 hour)
  Specific markers of inflammation measured in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Wendy E Ward, Ph.D., Principal Investigator — Brock University
Locations (1):
- Dr. Peter C. Fritz, Reconstructive Periodontics and Implant Surgery, Fonthill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No